CLINICAL TRIAL: NCT04943445
Title: A Single-arm, Multi-institutional, Phase 2 Study of a Pembrolizumab-based Organ Preservation Strategy for Locally Advanced Larynx Cancers
Brief Title: Study of a Pembrolizumab-based Organ Preservation Strategy for Locally Advanced Larynx Cancers
Acronym: SMART-KEY
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACOG 0720
Record Dates: First submitted 2021-06-16; First posted 2021-06-29 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Squamous Cell Carcinoma of Larynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Paclitaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment: Single Arm (Experimental): Induction chemo-immunotherapy:
  Carboplatin AUC of 6, paclitaxel 175 mg/m2, and pembrolizumab 200 mg, i.v. on day 1, every 21 days for 3 cycles. Patients without disease progression will proceed to the concurrent radioimmunotherapy phase of the trial.
  Concurrent radio-immunotherapy:
  Radiation therapy given concurrently with pembrolizumab 200 mg i.v. on day 1, every 21 days for 3 cycles. Patients without disease progression will proceed to the consolidation immunotherapy phase of the trial.
  Consolidation immunotherapy:
  Pembrolizumab 200 mg i.v. on day 1, every 21 days for 11 doses.
  Interventions: Drug: carboplatin AUC of 6, paclitaxel 175 mg/m2, and pembrolizumab 200 mg, i.v. on day 1, every 21 days for 3 cycles; Radiation: Concurrent radio-immunotherapy: radiation therapy given concurrently with pembrolizumab 200 mg i.v. on day 1, every 21 days for 3 cycles.; Drug: Consolidation immunotherapy: pembrolizumab 200 mg i.v. on day 1, every 21 days for 11 doses.

INTERVENTIONS:
Drug: carboplatin AUC of 6, paclitaxel 175 mg/m2, and pembrolizumab 200 mg, i.v. on day 1, every 21 days for 3 cycles — Patients without disease progression will proceed to the concurrent radioimmunotherapy phase of the trial.
Radiation: Concurrent radio-immunotherapy: radiation therapy given concurrently with pembrolizumab 200 mg i.v. on day 1, every 21 days for 3 cycles. — Patients without disease progression will proceed to the consolidation immunotherapy phase of the trial.
Drug: Consolidation immunotherapy: pembrolizumab 200 mg i.v. on day 1, every 21 days for 11 doses. — Consolidation immunotherapy

SUMMARY:
This a prospective, single-arm, multi-institutional, open label, phase 2 trial evaluating the effects of induction chemo-immunotherapy, followed by radioimmunotherapy, followed by consolidation immunotherapy in patients with locally advanced squamous cell carcinoma of the larynx who are candidates for organ preservation.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age on the day of signing informed consent
2. Histologically or cytologically confirmed new diagnosis of squamous cell carcinoma of the larynx (glottic or supraglottic).
3. Stages III, IVA, or IVB according to the AJCC (American Joint Cancer Committee) staging manual, 8th edition
4. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
5. Female participants:

   A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:
   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
6. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
7. If available, provision of an archived tumor tissue block (or at least 20 newly cut unstained slides) where such samples exist in a quantity sufficient to allow for analysis. A recent (≤3 months) tumor biopsy prior to treatment initiation is an optional requirement, provided that a biopsy procedure is technically feasible, and the procedure is not associated with unacceptable clinical risk. For patients without an available archival sample and who decline a new biopsy prior to study entry, enrolment without tissue provision will be allowed.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
9. Have adequate organ function

Exclusion Criteria:

1. Large volume T4 disease, defined as invasion through the cartilage or extension > 1 cm to the base of the tongue
2. T1 disease, defined as tumor limited to one subsite of the supraglottis or limited to the vocal cords, with normal vocal-cord mobility, according to the TNM staging system.
3. Contra indication, in the opinion of the treating physician, for radiotherapy, carboplatin or paclitaxel.
4. A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment initiation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

   a Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.

   b Creatinine clearance (CrCl) should be calculated per institutional standard. Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.
5. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).
6. Has received any prior systemic anti-cancer therapy for management of the participant's current cancer, including investigational agents prior to allocation.
7. Has received prior radiotherapy to the neck
8. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine.

   Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
9. Is currently participating in or has participated in a study of an investigational agent with anti-cancer activity or has used an investigational device within 4 weeks prior to the first dose of study intervention.
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
11. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.

    Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers
12. Has severe hypersensitivity (≥Grade 3) to pembrolizumab, carboplatin, paclitaxel and/or any of their excipients.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
14. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
15. Has an active infection requiring systemic therapy.
16. Has a known history of Human Immunodeficiency Virus (HIV) infection. Note: No HIV testing is required
17. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA qualitative detected) infection.

    Note: no testing for Hepatitis B and Hepatitis C is required
18. Has known active TB (Bacillus Tuberculosis).
19. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
22. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-10-16 (Estimated)

PRIMARY OUTCOMES:
Two-year laryngectomy-free survival | 24 months
  The primary efficacy endpoint is the two-year laryngectomy-free survival of patients with locally advanced larynx cancers treated with the study regimen. This endpoint combines assessment of both survival and larynx preservation and was used in the pivotal RTOG 91-11 study (12, 14), thus allowing for comparison with a historical control.

SECONDARY OUTCOMES:
Two-year larynx dysfunction-free survival | 24 months
  The secondary efficacy endpoint is two-year larynx dysfunction-free survival, which is a composite endpoint defined as the proportion of patients alive and without local recurrence and without lanryngoesophageal dysfunction. This endpoint reflects the necessity of evaluating not only survival with the larynx in place, but also laryngeal function, as stated in the recommendations by an international consensus panel (24). This endpoint was evaluated in the pivotal GORTEC 2000-01 trial (25, 26), thus allowing for comparisons with a historical control. Larynx dysfunction-free survival is also the primary endpoint of the ongoing, randomized, phase 3 trial GORTEC 2014-03, which will become a benchmark for larynx preservation studies in the near future. Predictive biomarkers of response survival will be evaluated as exploratory analysis.

CONTACTS AND LOCATIONS:
Overall Officials: William Nassib William Junior, Principal Investigator — Latin American Cooperative Oncology Group
Locations (10):
- Brazil (10):
  - CRIO - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - CPO - Centro de Pesquisa em Oncologia do Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor de Barretos, Barretos, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo
  - FUNFARME - Hospital de Base de São José do Rio Preto, São José do Rio Preto, São Paulo
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
  - ICESP - Instituto do Câncer do Estado de São Paulo, São Paulo
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo
  - A.C. Camargo Cancer Center, São Paulo